

## 1. PROTOCOL SYNOPSIS

| Investigational Product | SCS trial stimulator (Model 1000) |
|---|---|
| Title | A single-arm, open label, single center, prospective study of an ultra-high frequency spinal cord stimulation for treatment of chronic back pain or lower limb pain |
| Objectives | Primary: |
| | <ul> <li>To assess the analgesic effectiveness of ultra-high<br/>frequency spinal cord stimulation (as measured by<br/>VAS score compared to baseline)</li> </ul> |
| | <ul> <li>To evaluate safety of ultra-high frequency spinal cord<br/>stimulation by identifying the incidence rate of adverse<br/>events (AEs) and serious adverse events (SAEs)<br/>during the trial</li> </ul> |
| | Secondary: |
| | <ul> <li>The change from baseline in functionality using the<br/>BPI/ODI evaluations</li> </ul> |
| | <ul> <li>To determine the presence or absence of stimulation-<br/>induced paresthesia.</li> </ul> |
| | To assess the change of pain medication consumption |
| Indication | Pain control |
| Design | This study is a prospective, single-arm, open label, single center to confirm the effectiveness and safety of an ultra-high frequency spinal cord stimulation in patients with chronic back pain or lower limb pain. |
| Population | Inclusion criteria |
| | 1. Age ≧20 and ≦75 |
| | 2. Have a symptom of back or lower limb pain with a diagnosis related to spinal lesion, herniatic disc, nerve injury, stenosis, failed back surgery syndrome (FBSS), complex regional pain syndrome (CRPS) or ischemic lower limb pain and have pain history of <a href="mailto:&gt;6">6</a> months. |
| | 3. Have an average pain score >5 by Visual Analogue Scale |



(VAS) on inclusion.

- 4. Has failed to achieve adequate pain relief from prior pharmacologic treatments.
- 5. In the judgement of the investigator, the subject is an appropriate candidate for the trial procedure.
- 6. The subject is willing and able to comply with the procedure and requirements of this trial.
- 7. The participant is able to understand and provide informed consent, and has signed their written informed consent in accordance with IRB requirements.

## **Exclusion criteria**

- Have evidence of a mental or psychological condition that affects pain perception and has difficulty/disability performing objective pain assessment, or have previously failed mental or psychological assessments administered by a psychiatrist that may be deemed to indicate the subject's lack of suitability for participation in this study.
- 2. Subject has exhibited unstable pain condition within the past 30 days as interviewed by Investigator.
- 3. Be on anticoagulant medication with INR >1.5 or platelet count less than  $100,000/\mu L$ , peripheral vascular diseases (PVDs), visceral pain or uncontrolled Diabetes mellitus (DM).
- 4. Has had corticosteroid therapy at an intended site of stimulation within the past 30 days.
- 5. Pain medication(s) dosages(s) are not stable for at least 30 days at investigator's discretion.
- Currently has an active implantable device including ICD, pacemaker, spinal cord stimulator or intrathecal drug pump or subject requires magnetic resonance imaging (MRIs) or diathermy.
- 7. Have a current diagnosis of cancer with active symptoms.
- 8. Have a known terminal illness with life expectancy less than one year.
- 9. Have a systematic or local infection, which may increase study risk.



| MGE 13-5 | |
|---|---|
| | Currently has an indwelling device that may pose an increased risk of infection. |
| | 11. Be pregnant or breast feeding. |
| | 12. Have a medical history of drug or alcohol addiction within the past 2 years. |
| | 13. Participation in any investigational study in the last 30 days or current enrollment in any trial. |
| | 14. Be currently involved in an injury claim law suit or medically related litigation, including workers compensation. |
| | 15. Be a prisoner. |
| Sample Size | 10 evaluated subjects |
| Study Duration | 14 (+1) days |
| Efficacy Data | Primary endpoint: |
| | <ul> <li>Analgesic effectiveness of ultra-high frequency spinal<br/>cord stimulation (as measured by VAS score compare<br/>to baseline)</li> </ul> |
| | <ul> <li>Adverse event (AE) and serious AE (SAE) incidence<br/>rates during the trial</li> </ul> |
| | Secondary endpoints: |
| | Change in BPI/ODI compared to baseline |
| | Incidence of stimulation-induced paresthesia |
| | <ul> <li>Change in pain medication consumption, including<br/>Non-Steroidal Anti-Inflammatory Drugs (NSAIDs) and<br/>weak opioids, compared to baseline</li> </ul> |
| Statistical<br>Procedures | All data will be analyzed according to the full analysis set principle, including patients who received at least one dose of study treatment and had at least one follow-up evaluation regardless of their compliance with the protocol. Repeated measures analysis of variance (ANOVA) will be adopted to examine whether there are changes in VAS/BPI/ODI scores and pain medication consumption during the trail. The frequent endpoints in this study include AE, SAE and incidence of paresthesia of stimulation-induced. The incidence rates and their 95% confidence interval (CI) will be estimated. A Last Observation Carried Forward (LOCF) |

Protocol No.: PT1710001 Version 2.0, 05 Jan. 2018



method will be used to define endpoints if data is unavailable at the analysis time point; the last available measurement prior to the visit will be used to fill in the missing data. Interim analysis with Pocock-type group sequential plan will be undertaken for the likelihood of no merging trends and no reasonable chance of demonstrating benefit after 5 subjects are enrolled. The statistical significant level will be set at a two-tailed type 1 error of 0.05.

Protocol No.: PT1710001 CONFIDENTIAL

Version 2.0, 05 Jan. 2018